CLINICAL TRIAL: NCT00541632
Title: BacLite Rapid MRSA Clinical Performance
Status: Terminated | Type: Observational
Why Stopped: performance variability
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 010737
Record Dates: First submitted 2007-10-06; First posted 2007-10-10 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Methicillin Resistance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the performance of the 3M(TM) BacLite (TM) Rapid MRSA test system to traditional culture methods in detecting the presence of Methicillin Resistant Staphylococcus aureus (MRSA) directly from nasal samples.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older
* Subjects willing to document demographic characteristics
* Subjects willing to have their nose swabbed
* Subjects (or legal representative) willing to sign consent and authorization forms

Exclusion Criteria:

* Subjects who use Vicks Sinex Nasal spray or other nasal sprays
* Subjects with prescribed nasal medical devices where collecting samples may resent more than minimal risk to subjects
* Subjects having nasal prosthetics, jewelry or trauma to the nose or anything that may prevents sampling the anterior nares
* Investigator believes that subject is unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner E Bischoff, Principal Investigator — Wake Forest University
Locations (9):
- United States (9):
  - Denver Health Medical Center, Denver, Colorado
  - Atlanta Institute for Medical Research, Inc., Atlanta, Georgia
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio